CLINICAL TRIAL: NCT03679871
Title: Spiritual Assessment in Chronic Pain Patients: Construction and Validation of a Screening Tool in Health Care
Brief Title: Spiritual Assessment in Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Spiritual Care & Chronic Pain
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Chronic Pain; Spirituality
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaire validation (Other): 22-items questionnaire "Spiritual Resources and Distress"
  Interventions: Other: Questionnaire validation

INTERVENTIONS:
Other: Questionnaire validation — Participants will fill in the questionnaire "Spiritual Resources and Distress"plus additional questionnaires required for validation purposes. Three weeks later, a sub-sample will fill in the questionnaire one more time for consistency testing (test-retest)

SUMMARY:
The World Health Organization's (WHO) understanding of health(care) is incrementally incorporating the spiritual dimensions equivalent to the physical, psychological and social ones. Yet, it remains widely neglected in multi-modal, interprofessional chronic pain therapy. To support gaining access to chronic pain patients' spiritual needs and concerns within therapy, a screening tool has been constructed based on foregoing qualitative research and literature. The screening tool is to be validated with chronic pain patients in clinical settings.

DETAILED DESCRIPTION:
Addressing spiritual concerns and needs in chronic pain therapy is in line with the World Health Organization's (WHO) understanding of health(care) and would improve health care for this patient group. An applicable screening tool for chronic pain patients' spiritual concerns and needs must be empirically based. Based on preceding focus group interviews with patients and with health care professionals in various clinical settings and literature analysis, a screening tool has been constructed. This tool aims at supporting health care professionals as well as chronic pain patients in gaining access to spiritual concerns and needs for incorporation in multi-modal, interprofessional pain therapy. In this project the screening tools' psychometric properties will be tested with in five distinct clinical in- and out-patient settings.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient command of German language as assessed by local study coordinator
* Confirmed medical and/or nursing diagnosis of chronic pain
* Suffering pain for ≥ 6 months
* Pain intensity was≥ 5 on a 11-point numeric Rating scale (NRS; 0 = no pain, 10 = worst pain imaginable) during the last episode of pain

Exclusion Criteria:

* Life threatening diagnosis (e.g. cancer) that would introduce end-of-life topics as primary aspect
* Cognitive disorders that would impair participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Psychometric properties of "Spiritual Resources and Distress" questionnaire | 8 months
  Validity, internal consistency and stability of "Spiritual Resources and Distress" questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rufer, Prof., MD, Principal Investigator — University of Zurich
Locations (6):
- Switzerland (6):
  - Klinik SGM Langenthal, Langenthal, Canton of Bern
  - Schweizer Paraplegiker Zentrum, Zentrum für Schmerzmedizin, Nottwil, Canton of Lucerne
  - Zürcher RehaZentrum Davos, Davos, Kanton Graubünden
  - Arztpraxis Professor Sprott, Zurich
  - Universitätsspital Zürich, Institut für Anästhesiologie, Schmerzambulatorium, Zurich
  - Universitätsspital Zürich, Klinik für Konsiliarpsychiatrie und Psychosomatik, Zurich

REFERENCES:
- [Derived] Perrin J, Streeck N, Naef R, Rufer M, Peng-Keller S, Rettke H. Comparing perspectives: patients' and health care professionals' views on spiritual concerns and needs in chronic pain care - a qualitative study. BMC Health Serv Res. 2021 May 26;21(1):504. doi: 10.1186/s12913-021-06508-y. PMID 34039337